CLINICAL TRIAL: NCT01082224
Title: A Prospective, Multicenter Comparison of Multiphase Contrast-Enhanced CT and Multiphase Contrast-Enhanced MRI for Diagnosis of Hepatocellular Carcinoma and Liver Transplant Allocation
Brief Title: Contrast-Enhanced CT and MRI in Diagnosing and Staging Liver Cancer Using UNOS Policy
Acronym: ACRIN6690
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000667125; ACRIN-6690 (Other: CIP); U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — motexafin gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Waitlisted with HCC-Exception Points (Experimental): Participants undergo CT and MRI every 90 days for the trial with iodinated contrast dye and motexafin gadolinium, during liver transplant wait listing. Possible Eovist-enhanced MRI substudy participation
  Interventions: Drug: iodinated contrast dye; Drug: motexafin gadolinium; Other: Eovist-enhanced MRI

INTERVENTIONS:
Drug: iodinated contrast dye — iodinated Radiocontrast dye for imaging enhancement
  Other Names: iodinated radiographic dye
Drug: motexafin gadolinium — motexafin gadolinium
  Other Names: Xcytrin
Other: Eovist-enhanced MRI — A sub-study introduces the Eovist contrast agent for MRI scans at the same time points as the parent policy-assessment trial.

SUMMARY:
RATIONALE: Diagnostic procedures, such as contrast-enhanced CT scan and contrast-enhanced MRI, may help find liver cancer and find out how far the disease has spread.

PURPOSE: This clinical trial is studying contrast-enhanced CT scan and contrast-enhanced MRI in diagnosing and staging liver cancer in patients with chronic liver disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the sensitivity of multiphase contrast-enhanced CT scan to that of multiphase contrast-enhanced MRI using non-specific contrast agents for diagnosing hepatocellular carcinoma (HCC) in patients with chronic liver disease.

Secondary

* To compare the positive predictive value (PPV) of CT scan to that of MRI for diagnosing HCC.
* To compare the lesion-level sensitivity and PPV of CT scan and MRI as interpreted by radiologists at the respective transplant centers.
* To compare the sensitivity and specificity of multiphase contrast-enhanced CT scan vs MRI for diagnosing residual or recurrent HCC after local ablative therapy in patients listed for liver transplant.
* To determine the accuracy of imaging-based diagnosis and staging of HCC in clinical practice using the new Organ Procurement and Transplantation Network (OPTN) liver-imaging criteria compared with the reference standard of pathologic diagnosis and staging at the time of explantation.
* To explore whether the comparisons of sensitivity and PPV are affected by stratifying patients by AFP level (elevated vs normal). (Exploratory)

Tertiary

* To assess the sensitivity and PPV of MRI and CT interpreted at the participating sites on the basis of all available information and sequences and compare the sensitivity and PPV of the two modalities interpreted using the main study criterion. (Exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to AFP level (elevated vs normal).

Patients undergo CT scan with iodinated contrast agent and MRI with extracellular gadolinium contrast agent (both standard-of-care and study-related) at baseline and at 90-day intervals while on the liver transplant wait list.

After transplantation, the explanted liver will be analyzed for biomarkers and other studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Presence of ≥ 1 focal liver lesion(s) compatible with imaging diagnosis of stage II hepatocellular carcinoma (HCC) (Organ Procurement and Transplantation Network [OPTN] Class 5B liver lesion) on contrast-enhanced CT scan and/or contrast-enhanced MRI OR 2 or 3 focal liver lesions, each between > 1 and < 3 cm diameter, if each is compatible with imaging diagnosis of HCC on contrast-enhanced CT imaging and/or contrast-enhanced MRI

  * Imaging findings must be within the Milan criteria
* Listed on the regional OPTN/United Network for Organ Sharing (UNOS) liver transplant wait list with HCC-exception MELD points

  * Listed with the intent to undergo either deceased donor transplantation or live donor adult liver transplantation
* No evidence of any of the following:

  * Extrahepatic tumor
  * Unifocal tumor mass > 5 cm in diameter
  * Multifocal tumors ≥ 4 in number
  * Multiple (≤ 3) HCC with ≥ 1 tumor ≥ 3 cm in diameter

PATIENT CHARACTERISTICS:

* No renal failure, as determined by estimated GFR (eGFR) < 30 mL/min
* No renal insufficiency, as determined by eGFR 30-60 mL/min
* Not pregnant
* Negative pregnancy test
* Able to comply with breathing and other imaging-related instructions resulting in ability to obtain diagnostic-quality CT scan or MRI studies (OPTN Class 0)
* None of the following conditions that would make the patient unsuitable to undergo MRI with extracellular gadolinium-based contrast agent that does not have dominant hepatobiliary excretion:

  * Claustrophobia (unless alleviated with sedative treatment)
  * Presence of metallic objects or implanted medical devices in body per institutional safety standards
  * Sickle cell disease
  * Weight greater than that allowable by the MRI table
* None of the following conditions that would make the patient unsuitable to undergo CT scan with an iodinated contrast agent:

  * Iodinated contrast allergy
  * Weight greater than that allowable by the CT table
* No known allergy-like reaction to contrast media (iodinated or extracellular gadolinium that does not have dominant hepatobiliary excretion) or moderate or severe allergic reactions to one or more allergens as defined by the American College of Radiology and unwilling to undergo pre-treatment

PRIOR CONCURRENT THERAPY:

* No local ablative therapy to the liver before study enrollment
* No prior or concurrent sorafenib (or comparable antiangiogenic therapy)
* Patients planning to undergo local ablative therapy after transplant listing and study enrollment are eligible provided they undergo CT scan and MRI within 28-60 days after completing the last ablative therapy session
* Patients planning to receive transcatheter arterial chemoembolization (TACE) or combination therapy with TACE and thermal ablation are eligible provided they complete the entire treatment scheme per institutional standard of care before undergoing CT scan and MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2010-12; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of contrast-enhanced CT scan vs contrast-enhanced MRI for diagnosing hepatocellular carcinoma (HCC) | Within 90 Days Before Transplantation

SECONDARY OUTCOMES:
Positive predictive value (PPV) of CT scan vs MRI for diagnosing HCC | Within 90 Days Before Transplantation
Lesion-level sensitivity and PPV of contrast CT scan vs contrast MRI | Within 90 Days Before Transplantation
Sensitivity and specificity of multiphase contrast-enhanced CT scan vs MRI for diagnosing residual or recurrent HCC | Within 90 Days Before Transplantation
Accuracy of imaging-based diagnosis and staging of HCC in clinical practice using the new OPTN liver-imaging criteria compared with the reference standard of pathologic diagnosis and staging at the time of explantation | Within 90 Days Before Transplantation
Diagnostic value of sensitivity and PPV when patients are stratified by AFP level (elevated vs normal) | Within 90 Days Before Transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Wald, MD, PhD, Principal Investigator — Lahey Clinic Medical Center - Burlington
Locations (9):
- United States (9):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University, St. Louis, St Louis, Missouri
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Methodist Hospital for Liver Disease and Transplant, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan is available on-line at https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx

REFERENCES:
- [Result] Wald C, Nalesnik M, Pomfret EA, et al.: ACRIN 6690: can contemporary imaging reduce false-positive rate in liver transplant (LT) allocation? A multicenter comparison of CT and MRI for diagnosis of hepatocellular carcinoma (HCC). [Abstract] J Clin Oncol 29 (Suppl 15): A-TPS177, 2011.
- [Derived] Mitchell DG, Bruix J, Sherman M, Sirlin CB. LI-RADS (Liver Imaging Reporting and Data System): summary, discussion, and consensus of the LI-RADS Management Working Group and future directions. Hepatology. 2015 Mar;61(3):1056-65. doi: 10.1002/hep.27304. Epub 2014 Dec 12. PMID 25041904
- See also: ClinicalTrials.gov database — https://www.clinicaltrials.gov/ct2/show/NCT01082224?term=ACRIN-6690